CLINICAL TRIAL: NCT05969847
Title: Total Neoadjuvant Therapy With Split-course Hypofraction Radiotherapy Combined With CAPOX and Envafolimab Followed by Local Excision for Locally Advanced Very Low Rectal Cancer: an Open-label, Single-arm, Multi-center, Phase II Trial
Brief Title: Organ Preservation Following Enverolimab-based Total Neoadjuvant Therapy for Locally Advanced Very Low Rectal Cancer
Acronym: TRACE-LE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 池畔 (Other)
Responsible Party: Sponsor-Investigator, 池畔, Professor, Fujian Medical University Union Hospital
Organization: Fujian Medical University Union Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023XHYG0026-01
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Rectal Cancer
Keywords: Locally advanced very low rectal cancer; Total neoadjuvant therapy; Hypofraction radiotherapy; CAPOX; Envafolimab; Local excision
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX; envafolimab; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- split-course hypofraction radiotherapy plus CAPOX and Envafolimab followed by local excision (Experimental): Patients diagnosed with locally advanced very low rectal cancer were chosen to undergo a total neoadjuvant therapy (TNT) regimen. This regimen consisted of preoperative fractionated radiotherapy (5×7Gy) combined with 6 cycles of CAPOX chemotherapy and enverolimab.
  For patients who achieved clinical complete response (cCR) or near-clinical complete response (ncCR) after TNT, an organ-preserving strategy involving local full-thickness resection was implemented. Patients who achieve non-clinical complete response are subjected to traditional TME surgery.
  Interventions: Radiation: split-course hypofraction radiotherapy; Drug: CAPOX; Drug: Envafolimab; Procedure: Local excision

INTERVENTIONS:
Radiation: split-course hypofraction radiotherapy — After reaching a cumulative radiotherapy dose of 25Gy in the entire pelvic cavity (PTV1), the treatment field was subsequently narrowed to solely focus on the primary tumor (PTV2), with a total dose of 35Gy administered. All patients will undergo fractionated radiotherapy, following a regimen of 7Gy per fraction, delivered every 3 weeks for five cycles.
  Other Names: hypofraction radiotherapy
Drug: CAPOX — Drug: Oxaliplatin,130mg/m2，ivgtt，d1,for 6 cycles. Drug: Capecitabine,1000mg/m2，po，bid，d1-14, for 6 cycles.
  Other Names: Capecitabine+Oxaliplatin
Drug: Envafolimab — Envafolimab is administered by subcutaneous injection. The recommended dose is 300 mg per 3 weeks (Q3W) for 6 cycles.
  Other Names: KN035
Procedure: Local excision — Local full-thickness resection is employed for patients with clinical complete response (cCR) or near-clinical complete response (ncCR) following TNT.

SUMMARY:
Patients diagnosed with locally advanced very low rectal cancer were chosen to participate in a comprehensive neoadjuvant therapy (TNT) protocol. This treatment regimen consisted of preoperative fractionated radiotherapy (5×7Gy) combined with 6 cycles of CAPOX chemotherapy and enverolimab. For patients who achieved clinical complete response (cCR) or near-clinical complete response (ncCR) after undergoing TNT, an organ-preserving strategy involving local full-thickness resection was implemented.

DETAILED DESCRIPTION:
Locally advanced very low rectal cancer poses significant challenges in rectal cancer treatment. Presently, the prevailing approach in clinical practice involves neoadjuvant chemoradiotherapy in conjunction with total mesorectal excision (TME). Historically, abdominoperineal resection (APR) has been the conventional surgical procedure for managing locally advanced very low rectal cancer. However, the long-term presence of a colostomy following an abdominoperineal resection (APR) significantly impacts the quality of life for patients. Additionally, studies have revealed that 11.8-22% of rectal cancer patients who underwent APR after neoadjuvant chemoradiotherapy (nCRT) achieved a pathological complete response (pCR). Conversely, 11-52% of patients with pCR after nCRT for rectal cancer ultimately underwent APR surgery. Intersphincter resection (ISR) offers a highly beneficial surgical approach that preserves the anal sphincter, particularly for individuals with locally advanced very low rectal cancer. The patient's postoperative quality of life was significantly affected by severe low anterior resection syndrome (LARS), sexual dysfunction, and voiding dysfunction.

This study represents an exploratory phase II clinical trial in which patients diagnosed with locally advanced very low rectal cancer were chosen to undergo a total neoadjuvant therapy (TNT) regimen. This regimen consisted of preoperative fractionated radiotherapy (5×7Gy) combined with 6 cycles of CAPOX chemotherapy and enverolimab.

For patients who achieved clinical complete response (cCR) or near-clinical complete response (ncCR) after undergoing TNT, an organ-preserving strategy involving local full-thickness resection was implemented. Patients who achieve non-clinical complete response are subjected to traditional TME surgery.

This study aims to investigate the effectiveness and safety of organ preservation using the local resection approach in patients with locally advanced very low rectal cancer. By implementing this approach, the study aims to improve the quality of life for patients who achieve pathological complete response (pCR), thereby avoiding the need for conventional abdominoperineal resection (APR) and intersphincteric resection (ISR) procedures. Additionally, this study aims to address the issue of local regrowth associated with the "watch & wait" strategy and propose a novel treatment strategy for rectal-sparing surgery in patients with locally advanced very low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75.
2. Histopathology confirmed the rectal adenocarcinoma,cT3-4N0 or cT1-4N1-2. The tumor's lower margin ≤ 2cm from the anorectal ring's upper edge (based on MRI measurement).
3. Eastern tumor cooperation group (ECOG) status:0-2.
4. American Association of Anesthesiologists (ASA) status: I-III.
5. No previous systemic therapy, including chemotherapy, immunotherapy, or radiotherapy for rectal cancer.
6. No previous history of pelvic radiotherapy.
7. Sufficient organ function based on the following parameters:

   An absolute neutrophil count≥ 1.5 × 109 / L, a thrombocyte count ≥ 100 × 109/ L, a glomerular filtration rate (calculated using the Cockcroft-Gault formula) with a creatinine level ≤ 1.5 × ULN or a creatinine clearance > 50ml/min, and AST and ALT levels ≤ 2.5 × ULN or a total bilirubin level ≤ 1.5 × ULN.
8. Effective contraception during the study.
9. Patients are willing and able to comply with the protocol during the study period.
10. Patients with written informed consent

Exclusion Criteria:

1. Poorly differentiated adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, and adenocarcinoma developed from inflammatory bowel disease.
2. Metastasis to para-aortic, lateral, or inguinal lymph nodes has been identified.
3. Suspected distant metastasis in organs other than para-aortic, lateral, or inguinal lymph nodes is being considered.
4. Known hypersensitivity to platinum drugs or capecitabine.
5. Patients receiving concomitant treatment with drugs that interact with capecitabine or oxaliplatin (such as flucytosine, phenytoin, and warfarin).
6. According to the New York Heart Association (NYHA) classification, III or IV heart failure, and angina pectoris have occurred in the past six months.
7. Uncontrolled active infection or severe concomitant systemic disease.
8. Patients who need immunosuppressive therapy for organ transplantation.
9. Uncontrolled epilepsy or mental illness.
10. Pregnant or lactating female patients.
11. Non-compliance or researchers believe that the patient will not be able to complete the entire trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Organ preservation | 36 months
  The rectum is intact, owing to no radical total mesorectal excision (TME), curative (R0) salvage surgery by local excision (LE), and no permanent stoma (including a never reversed protective stoma or a stoma owing to toxicities and/or poor functional outcomes).

SECONDARY OUTCOMES:
ypT0-1 rate | 36 months
  The proportion of subjects with primary rectal cancer assessed by hematoxylin and eosin staining including no evidence of primary tumor (T0) or carcinoma in situ: intramucosal carcinoma (invading lamina propria, not infiltrating muscularis mucosa) (Tis) or tumor invading submucosa (T1) (ypT0-1 based on the latest UICC/AJCC staging system)
Pathological complete response (pCR) rate | 36 months
  Proportion of subjects with primary rectal cancer and all sampled lymph nodes who did not find any invasive carcinoma and high-grade intraepithelial neoplasia/severe dysplasia after assessment by hematoxylin and eosin staining (Judged as ypT0N0 stage according to the latest UICC/AJCC staging system)
Acute and late toxicity | 36 months
  Acute and late toxicity, Incidence of Treatment-Emergent Adverse Events assessment according to NCICTCAE V.5.0
Local recurrence rate | 36months
  The proportion of patients in all subjects within 3 years from the start of the surgery to detection of a tumor involving the bowel wall only that occurs after LE or TME
Local regional recurrence rate | 36 months
  The proportion of patients in all subjects within 3 years from the start of the surgery to detection of a tumor involving either the bowel wall, mesorectum, and/or pelvic organs that occurs after LE or TME
Disease-free survival | 36 months
  The proportion of patients in all subjects within 3 years from the start of the surgery to recurrence, distant metastsis, or death from any cause (whichever occurs first)
Quality of life-based on EORTC QLQ-C30 and EORTC QLQ-CR29 | baseline, 3 months, 12 months, 24 months, and 36 months after LE or TME
  Quality of life measured using EORTC QLQ-C30 and EORTC QLQ-CR29
Anorectal function | baseline, 3 months, 12 months, 24 months, and 36 months after LE or TME
  Anorectal function based on LARS score

CONTACTS AND LOCATIONS:
Overall Officials: Pan Chi, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Pan Chi, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No